CLINICAL TRIAL: NCT01177397
Title: A Phase 1/2, Multi-Center, Open-Label, Dose Finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of the mTOR Kinase Inhibitor CC-223 Administered Orally to Subjects With Advanced Solid Tumors, Non-Hodgkin Lymphoma, or Multiple Myeloma
Brief Title: Study to Assess Safety, Pharmacokinetics, and Efficacy of Oral CC-223 for Patients With Advanced Solid Tumors, Non-Hodgkin Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-223-ST-001
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2022-11-15 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Multiple Myeloma; Diffuse Large B-Cell Lymphoma; Glioblastoma Multiforme; Hepatocellular Carcinoma; Non-Small Cell Lung Cancer; Neuroendocrine Tumors of Non-Pancreatic Origin; Hormone Receptor-Positive Breast Cancer
Keywords: Advanced solid malignant neoplasms,Non-Hodgkin Lymphoma,; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Large B-Cell, Diffuse; Glioblastoma; Carcinoma, Hepatocellular; Carcinoma, Non-Small-Cell Lung | interventions — CC-223

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-223 (Experimental): All patients will receive CC-223, but serial patient groups will receive different dose levels in Phase 1. The number of groups will be determined by the number of dose levels required to establish dose-limiting toxicity.
  Interventions: Drug: CC-223

INTERVENTIONS:
Drug: CC-223 — Part A: (closed to enrollment) Dose level starts with 7.5mg daily taken by mouth in cycles of 28 days. Level increases for different patient cohorts in 100% or 50% increments until optimal dose level is established for further study. Treatment continues for as long as patient benefits (i.e., until disease progression or unacceptable toxicity). Part B: (closed to enrollment) Optimal dose is administered in 28 day cycles until disease progression.

SUMMARY:
The main purpose of this first human study with CC-223 is to assess the safety and action of a new class of experimental drug (dual mTOR inhibitors) in patients with advanced tumors unresponsive to standard therapies and to determine the appropriate dose and tumor type for later-stage clinical trials.

DETAILED DESCRIPTION:
Initially, patients will be treated with oral CC-223 for one month. During this time, various tests (involving blood and urine collections, ECGs, etc) will be performed. Those whose tumors stabilize or regress may continue receiving treatment for as long as they benefit from CC-223. Different dose levels of CC-223 will be tested in a dose-rising study design.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed advanced solid tumor, Non-Hodgkin Lymphoma or multiple myeloma
* Patients have not tolerated or progressed on standard therapy, and no further standard therapy is available
* Archival and screening tumor biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (solid tumors), 0-2 (hematologic malignancy)
* Adequate organ function

Exclusion Criteria:

* Prior systemic cancer-directed treatments or investigational drugs within 4 weeks or 5 half lives, whichever is shorter, prior to starting study drug or who have not recovered from side effects of such therapy. Subjects must have recovered from any effects of recent radiotherapy that might confound the safety evaluation of study drug
* Symptomatic brain metastases (prior Rx and stable metastases are OK)
* Acute or chronic liver or renal disease or pancreatitis
* Diarrhea ≥ Grade 2, impaired GI absorption
* Impaired cardiac function
* Diabetes requiring Rx, glucose >126 mg/dL, HbA1c ≥6.5%
* Peripheral neuropathy ≥ Grade 2
* Pulmonary fibrosis
* Known HIV infection
* Known chronic hepatitis B or C virus (HBV/HCV) infection, unless comorbidity in subjects with HCC
* Pregnant, inadequate contraception
* Most concurrent second malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2010-07-20 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (10):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Neuro-Oncology Program, Los Angeles, California
  - University of California, San Francisco Hellen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic Cancer Clinical Studies Unit, Rochester, Minnesota
  - Billings Clinic, Billings, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYU Cancer Institute - Bellevue Hospital, New York, New York
  - Sarah Cannon Research Institute Drug Development Unit, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas
- France (2):
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy Faculte de Medecine Paris Sud Service de pneumologie, Villejuif
- Spain (2):
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - UCL Cancer Institute, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: CC-223 7.5 mg: Participants received a single dose of 7.5 mg CC-223 on Day -1, then daily dosing of 7.5 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part A: CC-223 15 mg: Participants received a single dose of 15 mg CC-223 on Day -1, then daily dosing of 15 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part A: CC-223 30 mg: Participants received a single dose of 30 mg CC-223 on Day -1, then daily dosing of 30 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part A: CC-223 45 mg: Participants received a single dose of 45 mg CC-223 on Day -1, then daily dosing of 45 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part A: CC-223 60 mg: Participants received a single dose of 60 mg CC-223 on Day -1, then daily dosing of 60 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Non-small Cell Lung Cancer (NSCLC): Participants with NSCLC received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Glioblastoma Multiforme (GBM): Participants with GBM received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Hepatocellular Carcinoma (HCC): Participants with HCC received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Neuroendocrine Tumor (NET): Participants with NET received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Diffuse Large B-cell Lymphoma (DLBCL): Participants with DLBCL received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Multiple Myeloma (MM): Participants with MM received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
- Part B: Hormone Receptor Positive Breast Cancer (HRPBC): Participants with HRPBC received CC-223 at a starting dose of 45 mg/day (reduced to 30 mg/day after protocol Amendment 9) orally once a day in 28-day cycles for as long as they derived benefit from treatment as judged by the investigator.
Period: Overall Study
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Multiple Myeloma (MM) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC)
Started | 1 | 2 | 9 | 9 | 7 | 26 | 13 | 53 | 47 | 28 | 14 | 17
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 9 | 9 | 7 | 26 | 13 | 53 | 47 | 28 | 14 | 17
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 5 | 9 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0 | 12 | 1 | 14 | 8 | 6 | 3 | 7
Not completed — Disease progression | 1 | 2 | 5 | 5 | 4 | 10 | 10 | 21 | 18 | 12 | 10 | 8
Not completed — Other reasons | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 6 | 10 | 8 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Multiple Myeloma (MM) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC) | Total
Number analyzed (Participants) | 1 | 2 | 9 | 9 | 7 | 26 | 13 | 53 | 47 | 28 | 14 | 17 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant | 54.5 (10.61) | 53.8 (11.57) | 46.0 (12.86) | 49.9 (11.65) | 62.8 (10.72) | 55.6 (9.46) | 60.0 (11.41) | 62.6 (9.87) | 53.9 (14.51) | 60.4 (10.00) | 53.9 (7.79) | 58.2 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 6 | 5 | 6 | 12 | 5 | 10 | 28 | 11 | 6 | 17 | 108
  Male | 1 | 0 | 3 | 4 | 1 | 14 | 8 | 43 | 19 | 17 | 8 | 0 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 2 | 4 | 2 | 1 | 16
  Not Hispanic or Latino | 1 | 2 | 9 | 9 | 7 | 20 | 12 | 44 | 45 | 22 | 6 | 11 | 188
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 5 | 0 | 2 | 6 | 5 | 22
Race [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 10 | 2 | 0 | 0 | 1 | 20
  Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 0 | 0 | 9
  White | 1 | 2 | 7 | 7 | 6 | 20 | 12 | 31 | 43 | 24 | 8 | 10 | 171
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 4
  Missing | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 5 | 0 | 2 | 6 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose-limiting Toxicities
Description: A dose-limiting toxicity was defined as: - ≥ Grade 3 (per Common Terminology Criteria for Adverse Events [CTCAE] Version 4) clinically relevant adverse event (AE) or laboratory abnormality suspected to be related to CC-223 that commenced within 30 days of first dose, except alopecia, Grade 3 rash of the acneiform or maculopapular type for < 5 days, Grade 3 diarrhea or vomiting lasting < 72 hours, repeated occurrence of Grade 3 hyperuricaemia in subjects with Grade 3 hyperuricemia at baseline, hyperglycemia, hematologic and liver function test (LFT) abnormalities due to disease progression. - Grade 2 fasting hyperglycemia lasting > 14 days or ≥ Grade 3 lasting > 4 days despite optimal medical treatment. - Hematological toxicities including febrile neutropenia, Grade 4 neutropenia or thrombocytopenia for > 7 days, or Grade 3/4 thrombocytopenia with clinically significant bleeding. - Grade 4 LTFs - AE suspected to be CC-223 related necessitating dose reduction during cycle 1.
Time Frame: From first dose up to 30 days after first dose
Population: All treated participants in Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 9 | 9 | 7
Participants | 0 | 0 | 1 | 1 | 2

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of CC-223
Description: Cmax is defined as the maximum observed concentration (in plasma), obtained directly from the observed concentration versus time data. Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Cycle 1 Day 1: pre-dose, 0.5, 1, 1.5, 3, 5, 8, 24 and 48 hours post-dose and Day 15: pre-dose, 0.5, 1, 1.5, 3, 5, and 8 hours post-dose
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
ng/mL
  Day -1 | 45.8 (NA) — Coefficient of Variation not calculable because data were only collected for 1 participant. | 97.4 (57.5) | 188 (41.8) | 269 (65.7) | 319 (70.0)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 6 | 4
  Day 15 | 50.8 (NA) — Coefficient of Variation not calculable because data were only collected for 1 participant. | 92.0 (162.6) | 293 (38.8) | 417 (61.6) | 480 (88.9)

3. Primary Outcome: Time to Maximum Concentration (Tmax) of CC-223
Description: Tmax is defined as the time to Cmax, obtained directly from the observed concentration versus time data. Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: as for outcome 2
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
Hours
  Day -1/1 | 1.00 [1.00 to 1.00] | 1.25 [1.00 to 1.50] | 1.55 [1.00 to 3.20] | 3.00 [0.967 to 3.00] | 1.50 [1.00 to 5.00]
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 6 | 4
  Day 15 | 1.50 [1.50 to 1.50] | 2.00 [1.00 to 3.00] | 1.28 [0.500 to 3.03] | 1.63 [0.500 to 8.00] | 1.58 [1.00 to 3.00]

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUCt) for CC-223
Description: Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: Cycle 1 Day -1: pre-dose, 0.5, 1, 1.5, 3, 5, 8, 24 and 48 hours post-dose and Day 15: pre-dose, 0.5, 1, 1.5, 3, 5, and 8 hours post-dose
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
ng*h/mL
  Day -1/Day 1 | 318 (NA) — Insufficient data values to calculate coefficient of variation. | 347 (60.2) | 1204 (37.8) | 1493 (54.3) | 2080 (100.8)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 6 | 4
  Day 15 | 179 (NA) — Insufficient data values to calculate coefficient of variation. | 282 (100.7) | 1016 (39.2) | 1351 (45.0) | 1900 (93.5)

5. Primary Outcome: Area Under the Concentration Time-Curve From 0-24 Hours After a Dose (AUC0-24) for CC-223
Description: AUC0-24 is defined as the area under the concentration-time curve from Time 0 to 24 hours after a dose. Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: 0 to 24 hours post-dose on Day -1 and Day 15
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
ng*h/mL
  Day -1 | 319 (NA) — Insufficient data values to calculate coefficient of variation. | 379 (45.2) | 1144 (36.5) | 1497 (45.5) | 2031 (96.3)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 6 | 4
  Day 15 | 299 (NA) — Insufficient data values to calculate coefficient of variation. | 383 (88.8) | 1443 (41.4) | 2082 (29.3) | 2954 (106.2)

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf) For CC-223
Description: AUCinf is defined as the area under the concentration-time curve from Time 0 extrapolated to infinity. Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. AUCinf was not assessed following multiple dosing as the blood sampling schedule on Day 15 did not allow robust assessment of the terminal elimination rate constant.
Time Frame: as for outcome 2
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 8 | 6
ng*h/mL
  Day -1/1 | 353 (NA) — Insufficient data values to calculate coefficient of variation. | 378 (49.7) | 1234 (38.9) | 1694 (41.8) | 2074 (111.4)
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part A: Terminal Elimination Phase Half-Life (T1/2) of CC-223
Description: Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. T1/2 was not assessed following multiple dosing as the blood sampling schedule on Day 15 did not allow robust assessment of the terminal elimination rate constant.
Time Frame: Cycle 1 Day -1: pre-dose, 0.5, 1, 1.5, 3, 5, 8, 24 and 48 hours post-dose
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 8 | 6
Hours | 7.68 (NA) — Insufficient data values to calculate coefficient of variation. | 3.35 (54.1) | 5.57 (38.4) | 4.86 (25.9) | 5.64 (16.7)

8. Primary Outcome: Apparent Total Body Clearance (CL/F) of CC-223
Description: CL/F is defined as the apparent total body clearance when dosed orally, calculated as Dose/AUCinf. Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL.
Time Frame: as for outcome 2
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 8 | 6
L/h
  Day -1/1 | 21.2 (NA) — Insufficient data values to calculate coefficient of variation. | 39.7 (49.7) | 24.3 (38.9) | 26.6 (41.8) | 28.9 (111.4)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 6 | 4
  Day 15 | 25.1 (NA) — Insufficient data values to calculate coefficient of variation. | 39.2 (88.8) | 20.8 (41.4) | 21.6 (29.3) | 20.3 (106.2)

9. Primary Outcome: Apparent Volume of Distribution (Vz/F) of CC-223
Description: Plasma CC-223 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 1.00 ng/mL. VZ/F was not assessed following multiple dosing as the blood sampling schedule on Day 15 did not allow robust assessment of the terminal elimination rate constant.
Time Frame: Cycle 1 Day -1: pre-dose, 0.5, 1, 1.5, 3, 5, 8, 24 and 48 hours post-dose
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 8 | 6
L | 235 (NA) — Insufficient data values to calculate coefficient of variation. | 192 (3.70) | 195 (36.7) | 186 (27.1) | 236 (107.5)

10. Secondary Outcome: Part A: Percent Change From Baseline in Levels of Phosphorylated Ribosomal Protein S6 (pS6RP) in Stimulated B Cells
Description: Phosphorylated S6RP is a biomarker for inhibition of the mammalian target of rapamycin complex 1 (mTORC1). Phosphorylated S6RP was measured in stimulated B cells via flow cytometry. The raw measurements were expressed as median fluorescence intensity (MFI). MFI values were normalized against calibration beads using a linear regression transformation carried out on a log-log scale and reported as equivalent reference fluorophores (ERF). The biomarker evaluable population included all subjects who took at least one dose of study drug and had at least one non-missing pharmacodynamic (PD) assessment. Results were not available for the single subject treated in the 7.5-mg dose group and for one of the two subjects treated in the 15-mg dose group.
Time Frame: Cycle 1 Day -1: 3 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part A.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 0 | 1 | 6 | 8 | 7
Percent change
  Day -1 3 hours post-dose |  | -19.4 [-19.4 to -19.4] | -73.6 [-86.1 to -58.5] | -79.8 [-87.5 to -34.7] | -76.6 [-83.4 to -60.2]
  Day 15 1.5 hours post-dose: number analyzed (Participants) | 0 | 1 | 5 | 3 | 4
  Day 15 1.5 hours post-dose |  | 174.0 [174.0 to 174.0] | -59.0 [-77.5 to -41.3] | -80.5 [-84.6 to -80.0] | -69.3 [-86.2 to -61.7]

11. Secondary Outcome: Part A: Percent Change From Baseline in Levels of Phosphorylated Elongation I Initiation Binding Protein (p4E-BP1) in Stimulated T Cells
Description: Phosphorylated 4E-BP1 is a biomarker for inhibition of the mammalian target of rapamycin complex 1 (mTORC1). Phosphorylated 4E-BP1 was measured in stimulated T cells via flow cytometry. The raw measurements were expressed as median fluorescence intensity (MFI). MFI values were normalized against calibration beads using a linear regression transformation carried out on a log-log scale and reported as equivalent reference fluorophores (ERF). The biomarker evaluable population included all subjects who took at least one dose of study drug and had at least one non-missing pharmacodynamic (PD) assessment. Results were not available for the single subject treated in the 7.5-mg dose group and for one of the two subjects treated in the 15-mg dose group.
Time Frame: Cycle 1 Day -1: 3 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part A.
Measure: Median (Full Range); unit: Percent change in p4E-BP1
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 0 | 1 | 9 | 8 | 7
Percent change in p4E-BP1
  Day -1 3 hours post-dose |  | -20.7 [-20.7 to -20.7] | -44.0 [-65.1 to -28.7] | -55.7 [-71.2 to -26.4] | -44.3 [-63.7 to -1.0]
  Day 15 1.5 hours post-dose: number analyzed (Participants) | 0 | 1 | 6 | 4 | 4
  Day 15 1.5 hours post-dose |  | -14.4 [-14.4 to -14.4] | -61.1 [-92.8 to -44.5] | -54.8 [-61.8 to -34.4] | -46.4 [-69.8 to -26.3]

12. Secondary Outcome: Part A: Percent Change From Baseline in Levels of Phosphorylated Protein Kinase B (pAKT) in Stimulated Monocytes
Description: Phosphorylated AKT is a biomarker for inhibition of the mammalian target of rapamycin complex 2 (mTORC2). Phosphorylated AKT was measured in stimulated monocytes via flow cytometry. The raw measurements were expressed as median fluorescence intensity (MFI). MFI values were normalized against calibration beads using a linear regression transformation carried out on a log-log scale and reported as equivalent reference fluorophores (ERF). The biomarker evaluable population included all subjects who took at least one dose of study drug and had at least one non-missing pharmacodynamic (PD) assessment. Results were not available for the single subject treated in the 7.5-mg dose group and for one of the two subjects treated in the 15-mg dose group.
Time Frame: Cycle 1 Day -1: 3 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part A.
Measure: Median (Full Range); unit: Percent change in pAKT
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 0 | 1 | 9 | 8 | 7
Percent change in pAKT
  Day -1 3 hours post-dose |  | -26.9 [-26.9 to -26.9] | -56.5 [-72.2 to -31.7] | -59.7 [-74.6 to -23.0] | -48.4 [-53.6 to -26.7]
  Day 15 1.5 hours post-dose: number analyzed (Participants) | 0 | 1 | 6 | 3 | 4
  Day 15 1.5 hours post-dose |  | 58.3 [58.3 to 58.3] | -70.5 [-81.1 to -39.6] | -55.8 [-70.1 to -42.0] | -45.7 [-56.5 to -31.6]

13. Secondary Outcome: Part B: Percent Change From Baseline in p4E-BP1 in Monocytes by Tumor Cohort
Description: Phosphorylated 4E-BP1 is a biomarker for inhibition of the mammalian target of rapamycin complex 1 (mTORC1). Phosphorylated 4E-BP1 was measured in stimulated monocytes via flow cytometry. MFI values were determined and converted to molecules of equivalent fluorescence label (MEFL) by normalizing against calibration beads. The biomarker evaluable population included all subjects who took at least one dose of study drug and had at least one non-missing pharmacodynamic (PD) assessment. Data is reported by T-cell subsets known as clusters of differentiation (CD).
Time Frame: Cycle 1 Day 1: 1.5 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part B.
Measure: Median (Full Range); unit: Percent change in p4E-BP1
Arm/Group | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC) | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Multiple Myeloma (MM)
Number analyzed (Participants) | 10 | 44 | 34 | 15 | 6 | 18 | 3
Percent change in p4E-BP1
  Day 1,1.5 hours post-dose - CD3+: number analyzed (Participants) | 0 | 24 | 33 | 15 | 6 | 0 | 0
  Day 1,1.5 hours post-dose - CD3+ |  | -23.5 [-100.0 to 157.1] | -50.0 [-93.6 to 114.3] | -61.6 [-100.0 to 19.8] | -63.3 [-93.8 to 122.5] |  |
  Day 15, 1.5 hours post-dose - CD3+: number analyzed (Participants) | 0 | 18 | 22 | 10 | 5 | 0 | 0
  Day 15, 1.5 hours post-dose - CD3+ |  | -38.9 [-100.0 to 445.8] | -51.8 [-98.9 to 105.0] | -58.7 [-100.0 to 42.1] | -58.4 [-100.0 to 79.3] |  |
  Day 1,1.5 hours post-dose - CD14+: number analyzed (Participants) | 1 | 44 | 34 | 15 | 6 | 0 | 0
  Day 1,1.5 hours post-dose - CD14+ | -28.7 [-28.7 to -28.7] | -17.3 [-87.0 to 66.6] | -11.7 [-85.3 to 46.3] | -44.5 [-85.1 to 438.9] | -49.4 [-68.4 to 31.7] |  |
  Day 15, 1.5 hours post-dose - CD14+: number analyzed (Participants) | 1 | 19 | 23 | 10 | 5 | 0 | 0
  Day 15, 1.5 hours post-dose - CD14+ | -61.3 [-61.3 to -61.3] | -58.1 [-91.7 to 528.1] | -39.1 [-78.7 to 26.0] | -74.1 [-94.1 to 210.2] | -35.8 [-70.0 to 154.7] |  |
  Day 1,1.5 hours post-dose - CD19+: number analyzed (Participants) | 1 | 25 | 34 | 3 | 6 | 0 | 0
  Day 1,1.5 hours post-dose - CD19+ | -15.3 [-15.3 to -15.3] | -44.3 [-100.0 to 266.7] | -39.4 [-93.7 to 34.3] | -44.5 [-71.9 to -36.0] | -44.8 [-88.3 to 58.2] |  |
  Day 15, 1.5 hours post-dose - CD19+: number analyzed (Participants) | 1 | 18 | 23 | 3 | 5 | 0 | 0
  Day 15, 1.5 hours post-dose - CD19+ | -0.3 [-0.3 to -0.3] | -48.0 [-91.0 to 844.4] | -51.1 [-86.1 to 18.1] | -27.3 [-32.7 to -5.0] | -12.0 [-77.2 to 229.7] |  |
  Day 1,1.5 hours post-dose - CD91+: number analyzed (Participants) | 10 | 16 | 6 | 2 | 1 | 18 | 3
  Day 1,1.5 hours post-dose - CD91+ | -39.4 [-69.2 to 20.1] | -20.0 [-58.1 to 8.3] | -49.4 [-63.7 to -13.2] | -24.5 [-32.4 to -16.6] | -43.0 [-43.0 to -43.0] | -24.9 [-57.6 to 28.1] | -51.4 [-64.2 to -25.1]
  Day 15, 1.5 hours post-dose - CD91+: number analyzed (Participants) | 9 | 44 | 0 | 1 | 0 | 9 | 2
  Day 15, 1.5 hours post-dose - CD91+ | -22.4 [-53.7 to 151.3] | -24.7 [-39.7 to 16.8] |  | -6.9 [-6.9 to -6.9] |  | -24.8 [-38.4 to 77.5] | 19.6 [-7.9 to 47.2]

14. Secondary Outcome: Part B: Percent Change From Baseline in p4E-BP1 in Monocytes in the HCC and NET Cohorts by Dose
Description: as for outcome 13
Time Frame: Cycle 1 Day 1: 1.5 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part B.
Measure: Median (Full Range); unit: Percent change in p4E-BP1
Groups:
- HCC 30 mg: Participants with HCC received a daily dosing of 30 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- HCC 45 mg: Participants with HCC received a daily dosing of 45 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- NET 30 mg: Participants with NET received a daily dosing of 30 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- NET 45 mg: Participants with NET received a daily dosing of 45 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
Arm/Group | HCC 30 mg | HCC 45 mg | NET 30 mg | NET 45 mg
Number analyzed (Participants) | 20 | 6 | 21 | 13
Percent change in p4E-BP1
  Day 1 1.5 hours post-dose - CD3+: number analyzed (Participants) | 20 | 4 | 21 | 12
  Day 1 1.5 hours post-dose - CD3+ | -28.3 [-100.0 to 127.6] | 20.0 [-69.1 to 157.1] | -40.4 [-93.6 to 11.6] | -70.6 [-90.0 to 114.3]
  Day 15 1.5 hours post-dose - CD3+: number analyzed (Participants) | 15 | 3 | 15 | 7
  Day 15 1.5 hours post-dose - CD3+ | -34.0 [-100.0 to 445.8] | -52.8 [-62.6 to 52.4] | -39.7 [-95.7 to 33.8] | -70.2 [-98.9 to 105.0]
  Day 1 1.5 hours post-dose - CD14+ | -22.1 [-87.0 to 28.9] | 7.0 [-50.6 to 66.6] | -8.7 [-54.7 to 25.8] | -36.6 [-85.3 to 46.3]
  Day 15 1.5 hours post-dose - CD14+: number analyzed (Participants) | 15 | 4 | 15 | 8
  Day 15 1.5 hours post-dose - CD14+ | -58.1 [-91.7 to 528.1] | -28.4 [-67.5 to 111.6] | -25.6 [-78.7 to 26.0] | -47.4 [-68.3 to 23.2]

15. Secondary Outcome: Part B: Percent Change From Baseline in Levels of pAKT in Monocytes by Tumor Cohort
Description: Phosphorylated AKT is a biomarker for inhibition of the mammalian target of rapamycin complex 2 (mTORC2). Phosphorylated AKT was measured in stimulated monocytes via flow cytometry. MFI values were determined and converted to molecules of equivalent fluorescence label (MEFL) by normalizing against calibration beads. The biomarker evaluable population included all subjects who took at least one dose of study drug and had at least one non-missing pharmacodynamic (PD) assessment.
Time Frame: Cycle 1 Day 1: 1.5 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part B.
Measure: Median (Full Range); unit: Percent change in pAKT
Arm/Group | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Multiple Myeloma (MM) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC)
Number analyzed (Participants) | 16 | 8 | 16 | 4 | 2 | 4 | 1
Percent change in pAKT
  Day 1 1.5 hours post-dose | -68.1 [-86.5 to 43.9] | -28.0 [-73.0 to 130.1] | -55.5 [-86.2 to 27.1] | -70.3 [-83.7 to -51.2] | -54.3 [-89.0 to -19.6] | -78.8 [-86.2 to -27.1] | -53.8 [-53.8 to -53.8]
  Day 15 1.5 hours post-dose: number analyzed (Participants) | 8 | 8 | 7 | 1 | 1 | 2 | 0
  Day 15 1.5 hours post-dose | -76.1 [-93.0 to -27.5] | -34.1 [-89.8 to 48.6] | -84.1 [-87.7 to -19.5] | -52.2 [-52.2 to -52.2] | -88.6 [-88.6 to -88.6] | -52.9 [-77.5 to -28.2] |

16. Secondary Outcome: Part B: Percent Change From Baseline in Levels of pAKT in Monocytes in the HCC and NET Cohorts by Dose
Description: as for outcome 15
Time Frame: Cycle 1 Day 1: 1.5 hours post-dose and Day 15: 1.5 hours post-dose
Population: All biomarker evaluable participants who received treatment in Part B.
Measure: Median (Full Range); unit: Percent change in pAKT
Groups:
- HCC 30mg: Participants with HCC received a daily dosing of 30 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- HCC 45mg: Participants with HCC received a daily dosing of 45 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- NET 30mg: Participants with NET received a daily dosing of 30 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
- NET 45mg: Participants with NET received a daily dosing of 45 mg CC-223 for 28 days beginning on Day 1. Participants received subsequent cycles consisting of 28-day continuous dosing without rest between cycles for as long as they derived benefit from treatment as judged by the investigator.
Arm/Group | HCC 30mg | HCC 45mg | NET 30mg | NET 45mg
Number analyzed (Participants) | 0 | 16 | 0 | 4
Percent change in pAKT
  Day 1 1.5 hours post-dose |  | -55.5 [-86.2 to 27.1] |  | -70.3 [-83.7 to -51.2]
  Day 15 1.5 hours post-dose: number analyzed (Participants) | 0 | 7 | 0 | 1
  Day 15 1.5 hours post-dose |  | -84.1 [-87.7 to -19.5] |  | -52.2 [-52.2 to -52.2]

17. Secondary Outcome: Part B: Percent Change From Baseline in pS6RP Levels in Tumor Tissue by Tumor Type
Description: Tumor tissue biopsies were performed at Baseline and on Day 15 3 hours post dose. Levels of pS6RP were quantified using immunohistochemical (IHC) methods.
Time Frame: Up to Cycle 1 Day 15 3 hours post dose
Population: All biomarker evaluable participants who received treatment in Part B.
Measure: Median (Full Range); unit: Percent change in pS6RP
Arm/Group | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Multiple Myeloma (MM) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC)
Number analyzed (Participants) | 6 | 1 | 3 | 1 | 9 | 0 | 3
Percent change in pS6RP | 22 (-37) [-37 to 66] | -36 (-36) [-36 to -36] | -19 (-37) [-37 to 24] | -30 (-30) [-30 to -30] | -21 (-43) [-43 to 12] |  | -15 (-17) [-17 to 6]

18. Secondary Outcome: Part A: Overall Response Rate
Description: Tumor response was based on Investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for solid tumors (NSCLC, HCC, NET, and HRPBC), and the International Working Group Criteria (IWC) for DLBCL. Overall Response Rate is defined as the percentage of participants with a best overall response of complete response or partial response. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. In Part A, participants with MM and participants with GBM were not evaluated for tumor response.
Time Frame: From first dose up to tumor response (approximately 11 months)
Population: Participants who received treatment in Part A
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 9 | 9 | 7
Percentage of participants | 0 | 0 [NA to NA] — Lower and upper limit not calculated due to insufficient number of events | 11.1 [0.6 to 42.9] | 0 [NA to NA] — Lower and upper limit not calculated due to insufficient number of events | 0 [NA to NA] — Lower and upper limit not calculated due to insufficient number of events

19. Secondary Outcome: Part B: Overall Response Rate
Description: Tumor response was based on Investigator assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for solid tumors (NSCLC, HCC, NET, and HRPBC), International Working Group Criteria (IWC) for DLBCL, and the International Myeloma Working Group (IMWG) criteria for MM. For GBM, Responses Assessment for Neuro-Oncology Working Group (RANO) criteria were used for tumor response, using the post resection MRI scan as the baseline. Overall Response Rate is defined as the percentage of participants with a best overall response of complete response or partial response. Complete response is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to tumor response (approximately 36 months)
Population: Participants who received treatment in Part B reported by tumor cohort
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Multiple Myeloma (MM) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC)
Number analyzed (Participants) | 26 | 13 | 53 | 47 | 28 | 14 | 17
Percentage of participants | 3.8 [0.1 to 19.6] | 0 [NA to NA] — Lower and upper limit not calculated due to insufficient number of events | 5.7 [1.2 to 15.7] | 6.4 [1.3 to 17.5] | 10.7 [2.3 to 28.2] | 0 [NA to NA] — Lower and upper limit not calculated due to insufficient number of events | 11.8 [1.5 to 36.4]

20. Secondary Outcome: Maximum Observed Concentration (Cmax) of Metabolite M1
Description: Cmax is defined as the maximum observed concentration (in plasma), obtained directly from the observed concentration versus time data. Plasma metabolite M1 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 10.0 ng/mL.
Time Frame: as for outcome 4
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
ng/mL
  Day -1 | 143 (NA) — Insufficient data values to calculate coefficient of variation. | 284 (64.6) | 729 (40.3) | 1002 (37.2) | 1174 (86.0)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 7 | 5
  Day 15 | 363 (NA) — Insufficient data values to calculate coefficient of variation. | 357 (139.8) | 1681 (34.5) | 2061 (23.1) | 1946 (78.9)

21. Secondary Outcome: Time to Maximum Concentration (Tmax) of Metabolite M1
Description: Tmax is defined as the time to Cmax, obtained directly from the observed concentration versus time data. Plasma metabolite M1 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 10.0 ng/mL.
Time Frame: as for outcome 4
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
Hours
  Day 1 | 8.00 [8.00 to 8.00] | 2.28 [1.50 to 3.05] | 6.51 [1.50 to 8.00] | 5.00 [1.60 to 8.00] | 5.00 [1.67 to 8.00]
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 7 | 5
  Day 15 | 1.50 [1.50 to 1.50] | 3.25 [1.50 to 5.00] | 1.58 [1.00 to 3.03] | 1.71 [0.00 to 3.20] | 3.00 [0.00 to 5.00]

22. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUCt) for Metabolite M1
Description: AUCt is defined as the area under the concentration-time curve from Time 0 to the time of the last quantifiable concentration. Plasma metabolite M1 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 10.0 ng/mL.
Time Frame: as for outcome 4
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
ng*h/mL
  Day 1 | 4583 (NA) — Insufficient data values to calculate coefficient of variation. | 3788 (121.2) | 18964 (45.1) | 19938 (30.1) | 23702 (98.1)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 7 | 5
  Day 15 | 6401 (NA) — Insufficient data values to calculate coefficient of variation. | 4388 (133.8) | 27389 (48.5) | 30823 (38.3) | 33070 (101.6)

23. Secondary Outcome: Area Under the Concentration Time-Curve From 0-24 Hours After a Dose (AUC0-24) for Metabolite M1
Description: AUC0-24 is defined as the area under the concentration-time curve from Time 0 to 24 hours after a dose. Plasma metabolite M1 was measured using validated chiral liquid chromatography-mass spectrometry methods (LC-MS/MS). The lower limit of quantification (LLOQ) in plasma was 10.0 ng/mL.
Time Frame: 0 to 24 hours post-dose on Day -1 and Day 15
Population: All treated participants with available pharmacokinetic data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg
Number analyzed (Participants) | 1 | 2 | 8 | 9 | 7
ng*h/mL
  Day 1 | 2712 (NA) — Insufficient data values to calculate coefficient of variation. | 3207 (82.5) | 12328 (39.4) | 14107 (26.9) | 16926 (89.2)
  Day 15: number analyzed (Participants) | 1 | 2 | 6 | 7 | 5
  Day 15 | 6401 (NA) — Insufficient data values to calculate coefficient of variation. | 4388 (133.8) | 27389 (48.5) | 30823 (38.3) | 33070 (101.6)

24. Primary Outcome: Part B: Progression Free Survival (PFS) Rate at 6 Months for GBM Participants
Description: Progression free survival rate of GBM participants at 6 months is defined as the percentage of participants without progressive disease per Evaluation Criteria in Solid Tumors (RECIST) 1.1 6 months after starting study treatment. Progressive disease is defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: From first dose to 6 months
Population: All treated participants in Part B with GBM without progression per RECIST 1.0 at 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Glioblastoma Multiforme (GBM)
Number analyzed (Participants) | 13
Percentage of participants | 0 [NA to NA] — Lower and upper limit not reached to insufficient number of events

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From first dose through the course of the trial (up to approximately 6 years). Part A SAEs and AEs: From first dose to 100 days post last dose (up to approximately 14 months). Part B SAEs and AEs: From first dose to 100 days post last dose (up to approximately 49 months).
Description: Although the protocol stated Part B participants would begin treatment at the MTD determined by Part A (45 mg), the conduct of Part B permitted participants to stay in the study even though they had many dose reductions and dosing interruptions. Dosing/exposure for participants varied greatly and there were few participants which remained at any given dose for most of the study. Due to this, there was no analysis of Part B data available according to dose.
Arm/Group | Part A: CC-223 7.5 mg | Part A: CC-223 15 mg | Part A: CC-223 30 mg | Part A: CC-223 45 mg | Part A: CC-223 60 mg | Part B: Non-small Cell Lung Cancer (NSCLC) | Part B: Glioblastoma Multiforme (GBM) | Part B: Hepatocellular Carcinoma (HCC) | Part B: Neuroendocrine Tumor (NET) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) | Part B: Multiple Myeloma (MM) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 2/9 | 3/9 | 1/7 | 10/26 | 3/13 | 24/53 | 2/47 | 5/28 | 2/14 | 4/17
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 4/9 | 4/9 | 2/7 | 15/26 | 6/13 | 29/53 | 23/47 | 17/28 | 6/14 | 11/17
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 8/9 | 9/9 | 7/7 | 26/26 | 13/13 | 53/53 | 47/47 | 28/28 | 14/14 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: CC-223 7.5 mg (N=1) | Part A: CC-223 15 mg (N=2) | Part A: CC-223 30 mg (N=9) | Part A: CC-223 45 mg (N=9) | Part A: CC-223 60 mg (N=7) | Part B: Non-small Cell Lung Cancer (NSCLC) (N=26) | Part B: Glioblastoma Multiforme (GBM) (N=13) | Part B: Hepatocellular Carcinoma (HCC) (N=53) | Part B: Neuroendocrine Tumor (NET) (N=47) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) (N=28) | Part B: Multiple Myeloma (MM) (N=14) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC) (N=17)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perihepatic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusional disorder, persecutory type (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: CC-223 7.5 mg (N=1) | Part A: CC-223 15 mg (N=2) | Part A: CC-223 30 mg (N=9) | Part A: CC-223 45 mg (N=9) | Part A: CC-223 60 mg (N=7) | Part B: Non-small Cell Lung Cancer (NSCLC) (N=26) | Part B: Glioblastoma Multiforme (GBM) (N=13) | Part B: Hepatocellular Carcinoma (HCC) (N=53) | Part B: Neuroendocrine Tumor (NET) (N=47) | Part B: Diffuse Large B-cell Lymphoma (DLBCL) (N=28) | Part B: Multiple Myeloma (MM) (N=14) | Part B: Hormone Receptor Positive Breast Cancer (HRPBC) (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (12) | 0 (0) | 5 (5) | 3 (3) | 8 (9) | 7 (24) | 5 (10)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 3 (8) | 6 (12) | 4 (18) | 3 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 4 (7) | 2 (2) | 16 (30) | 5 (14) | 11 (23) | 7 (29) | 6 (9)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scintillating scotoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 2 (3) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 14 (20) | 15 (24) | 5 (8) | 0 (0) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 1 (1)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 3 (5)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (9) | 0 (0) | 0 (0) | 2 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 9 (10) | 0 (0) | 12 (13) | 9 (10) | 8 (10) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 5 (5) | 5 (6) | 16 (41) | 5 (6) | 32 (55) | 36 (138) | 17 (29) | 7 (9) | 11 (21)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 4 (4) | 9 (10) | 4 (5) | 3 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (2)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 3 (3)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 6 (6) | 3 (4) | 16 (28) | 9 (13) | 27 (40) | 22 (34) | 13 (16) | 7 (12) | 12 (21)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 13 (20) | 3 (3) | 15 (30) | 25 (52) | 5 (6) | 9 (10) | 8 (16)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (5) | 6 (7) | 13 (27) | 2 (3) | 15 (21) | 11 (14) | 9 (11) | 8 (11) | 8 (13)
Asthenia (General disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 15 (37) | 1 (1) | 14 (23) | 18 (31) | 7 (10) | 8 (13) | 5 (14)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 2 (2) | 6 (7) | 5 (7) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2) | 4 (7) | 6 (8) | 7 (10) | 17 (38) | 4 (7) | 32 (63) | 33 (68) | 11 (17) | 2 (2) | 8 (25)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 10 (10) | 0 (0) | 0 (0) | 1 (1)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 5 (9) | 0 (0) | 1 (4) | 7 (11) | 6 (12) | 4 (4) | 0 (0) | 4 (8)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (7) | 0 (0) | 1 (1) | 2 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 5 (6) | 2 (4) | 11 (14) | 14 (30) | 2 (2) | 0 (0) | 3 (4)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 4 (6) | 5 (9) | 4 (4) | 13 (18) | 8 (14) | 3 (3) | 1 (1) | 2 (3)
Thirst decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 3 (4) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 7 (10) | 9 (16) | 2 (2) | 1 (1) | 3 (3)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 16 (22) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 23 (46) | 5 (9) | 2 (3) | 2 (2) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 12 (23) | 3 (7) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (12) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 3 (6) | 3 (6) | 0 (0) | 3 (11) | 3 (4)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 9 (22) | 1 (2) | 12 (35) | 12 (22) | 5 (7) | 6 (12) | 3 (7)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (6) | 1 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulse pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tandem gait test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 9 (12) | 0 (0) | 17 (24) | 7 (10) | 5 (5) | 3 (3) | 4 (4)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cell death (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (6) | 4 (6) | 2 (2) | 19 (34) | 3 (3) | 34 (52) | 21 (33) | 15 (22) | 6 (11) | 11 (22)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 10 (11) | 1 (1) | 13 (18) | 14 (30) | 2 (2) | 1 (1) | 4 (8)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (8) | 4 (11) | 3 (5) | 14 (37) | 3 (3) | 32 (75) | 15 (38) | 10 (22) | 8 (16) | 7 (20)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 3 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 2 (5) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (10) | 2 (3) | 8 (12) | 11 (18) | 10 (16) | 1 (1) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 5 (7) | 0 (0) | 3 (5) | 0 (0) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (16) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (12) | 2 (3) | 11 (28) | 3 (3) | 5 (9) | 2 (4) | 3 (5)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 4 (5) | 6 (11) | 0 (0) | 1 (2) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 5 (6) | 0 (0) | 4 (4) | 10 (12) | 4 (4) | 4 (4) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 2 (2) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (6) | 3 (4) | 0 (0) | 4 (4)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 6 (8) | 3 (4) | 7 (7) | 13 (17) | 3 (3) | 1 (1) | 2 (3)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (5) | 1 (1) | 11 (14) | 8 (13) | 0 (0) | 1 (1) | 2 (2)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 5 (10) | 11 (11) | 8 (8) | 6 (7) | 3 (3) | 5 (5)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incoherent (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (5) | 3 (3) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Quadrantanopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Upper motor neurone lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White matter lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anhedonia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 3 (4) | 3 (3) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (15) | 5 (7) | 0 (0) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 2 (7) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (2) | 2 (2) | 5 (7) | 0 (0) | 8 (11) | 9 (12) | 0 (0) | 0 (0) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 2 (2) | 15 (29) | 1 (3) | 10 (13) | 10 (15) | 3 (3) | 1 (1) | 7 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (9) | 0 (0) | 8 (13) | 8 (8) | 0 (0) | 2 (2) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 9 (21) | 1 (1) | 18 (41) | 21 (47) | 5 (5) | 2 (2) | 6 (8)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (4) | 3 (4) | 8 (13) | 4 (5) | 12 (18) | 18 (39) | 5 (6) | 3 (6) | 4 (19)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 7 (26) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (8) | 2 (2) | 7 (22) | 12 (22) | 2 (2) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (7) | 3 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (15) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 5 (6) | 4 (4) | 2 (2) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.